CLINICAL TRIAL: NCT00003714
Title: Phase II Trial of Pyrazoloacridine (PZA) in Previously Untreated Hepatocellular Carcinoma (HCC) Patients
Brief Title: Chemotherapy in Treating Patients With Unresectable Primary or Metastatic Kidney Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM98-107; P30CA016672 (NIH); U01CA070172 (NIH); MDA-DM-98107 (Other: UT MD Anderson Cancer Center); NCI-T98-0031; CDR0000066822 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-09-14 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Liver Cancer; Metastatic Cancer
Keywords: localized unresectable adult primary liver cancer; advanced adult primary liver cancer; adult primary hepatocellular carcinoma; liver metastases
MeSH Terms: conditions — Liver Neoplasms; Neoplasm Metastasis; Carcinoma, Hepatocellular | interventions — NSC 366140

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pyrazoloacridine (Experimental)
  Interventions: Drug: Pyrazoloacridine

INTERVENTIONS:
Drug: Pyrazoloacridine — IV (by vein) over 3 hours every 3 weeks
  Other Names: PZA

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of pyrazoloacridine in treating patients who have unresectable primary or metastatic kidney cancer that has not been previously treated.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate, duration, and survival in previously untreated patients with hepatocellular carcinoma treated with pyrazoloacridine (PZA). II. Determine the nature, degree, and duration of toxic effects of PZA in these patients.

OUTLINE: Patients receive pyrazoloacridine IV over 3 hours every 3 weeks. The minimum treatment period is 2 courses with tumor restaging at 6 weeks. Patients with complete remission (CR) or partial remission (PR) may continue on treatment until refractory (PR) or for at least 3 additional courses (CR). Patients with stable disease continue on therapy for at least 2 more courses. Patients are followed until death.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study within 24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven unresectable primary or metastatic hepatocellular carcinoma Measurable disease by CT or MRI scan No tense ascites Brain metastases allowed with proper treatment

PATIENT CHARACTERISTICS: Age: Not specified Performance status: Karnofsky 70-100% Zubrod 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Albumin at least 3 g/dL Alkaline phosphatase no greater than 3 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL Other: Not pregnant or nursing Fertile patients must use effective contraception No significant infection Peripheral neurologic toxicity limited to paresthesia and decreased vibratory sense without motor weakness allowed Constipation managed with laxatives without evidence of bowel obstruction allowed No psychological disorders including delirium, confusion, suicidal ideation, or untreated depression

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: Prior palliative radiotherapy allowed At least 3 weeks since prior radiotherapy and recovered Surgery: Recovered from any prior surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Patient Response | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Z. Patt, MD, Study Chair — M.D. Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org